CLINICAL TRIAL: NCT06255964
Title: A Phase I/II Clincal Trial of Intravesical IAP0971 in Combination With Bacillus Calmette Guerin (BCG) in Patients With BCG Unresponsive High Risk Non-Muscular Invasive Bladder Cancer (NMIBC)
Brief Title: A Study of IAP0971 in Combination With Bacillus Calmette Guerin in High Risk Non-muscular Invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IAP0971-201
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase Ia study (Other): Phase Ia study: for adults with BCG treatment failure or intolerance to BCG, high-risk non muscle invasive bladder cancerPatient, evaluate the safety and tolerability of IAP0971 monotherapy bladder infusion, and determine dose limiting toxicity and/or phase II recommended dose.
  Interventions: Drug: IAP0971
- Phase Ib study (Experimental): Phase Ib study:To evaluate the safety and tolerability of intravesical IAP0971 in combination with BCG in patients with BCG unresponsive high risk non-muscle invasive bladder cancer, and to determine the DLT and RP2D.
  Interventions: Combination Product: IAP0971＋BCG
- Phase II study (Experimental): Phase II study:To evaluate the efficacy of intravesical IAP0971 in combination with BCG in patients with BCG unresponsive high risk NMIBC using RP2D as determined in the phase I study.
  Interventions: Combination Product: IAP0971＋BCG

INTERVENTIONS:
Drug: IAP0971 — Induction period (6 weeks): IAP0971 single drug bladder infusion, once a week;Maintenance period: IAP0971 single drug bladder infusion, performed at 3, 6, 12, 18, and 24 months, once a week, for 3 consecutive times
  Arms: Phase Ia study
Combination Product: IAP0971＋BCG — Induction period (6 weeks): IAP0971 combined with BCG,Bladder perfusion, once a week;Maintenance period: IAP0971 combined with BCG bladder perfusion,Maintain at months 3, 6, 12, 18, and 24Perfusion, once a week, three times in a row.
  Arms: Phase Ib study
Combination Product: IAP0971＋BCG — Induction period (6 weeks): IAP0971 combined with BCG,Bladder perfusion, once a week;Maintenance period: IAP0971 combined with BCG bladder irrigationNote, progress at months 3, 6, 12, 18, and 24Perform maintenance perfusion once a week, three times in a row.
  Arms: Phase II study

SUMMARY:
The efficacy and safety of IAP0971 single drug or combined with BCG intravesical instillation in the treatment of high-risk non muscle invasive bladder cancer with BCG treatment failure.

DETAILED DESCRIPTION:
Phase Ia study: for adults with BCG treatment failure or intolerance to BCG, high-risk non muscle invasive bladder cancerPatient, evaluate the safety and tolerability of IAP0971 monotherapy bladder infusion, and determine dose limiting toxicity and/or phase II recommended dose.

Phase Ib study:To evaluate the safety and tolerability of intravesical IAP0971 in combination with BCG in patients with BCG unresponsive high risk non-muscle invasive bladder cancer, and to determine the DLT and RP2D.

Phase II study:To evaluate the efficacy of intravesical IAP0971 in combination with BCG in patients with BCG unresponsive high risk NMIBC using RP2D as determined in the phase I study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years on the day of signing informed consent form.
2. Patients who have NMIBC which is confirmed by cystoscopy, urine cytology and histopathology examination within 12 weeks prior to the first dose, and is classified as high risk according to the Guideline of Non-muscle Invasive Bladder Cancer issued by European Association of Urology (EAU) (version 2021)
3. CIS patients must have CIS on the tumor sample from the most recent cystoscopy/TURBT.
4. Patients who have papillary tumors (Ta and T1), a complete TURBT must have been performed, as characterized by:

   -Attainment of a visually complete resection of all papillary tumors (Ta and T1);

   -Residual CIS, therefore not amenable to complete transurethral resection is acceptable;
   * The most recent cystoscopy/TURBT must have been performed within 12 weeks prior to the first dose.
5. Patients who have received and failed BCG intravesical instillation therapy prior to enrollment and are ineligible for radical cystectomy or elect not to undergo the procedure.

   Failure of BCG therapy including: BCG refractory tumor, BCG relapsing tumor, BCG unresponsive tumor
6. Patients who have elected not to undergo the radical cystectomy or are ineligible for the procedure on the investigator's judgment. The reasons for ineligible or refusal of radical cystectomy should be discussed with the patient as part of the informed consent and should be documented on the appropriate case report form. Ineligibility factors for radical cystectomy include, but are not limited to:

   -Patients have cardiovascular disease (e.g., recent acute coronary syndrome, cardiac arrhythmias, heart failure);

   -Patients have chronic obstructive pulmonary disease that would preclude a safe surgical procedure, as determined by the treating surgeon;

   -Patients have undergone major abdominal and pelvic surgery that would preclude a safe surgical procedure, as determined by the treating surgeon.
7. Patients who have a performance status of 0 or 1 on the ECOG performance scale
8. Adequate organ function during the screening period, include:

   -Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;

   -Hemoglobin (Hgb) ≥ 80 g/L;

   -Platelets (PLT) ≥ 100 × 10^9/L;

   -ALT and AST ≤ 2.5 × ULN, or ≤ 5.0 × ULN for subject with liver metastases;
   * Total bilirubin (TBIL) ≤ 1.5×ULN;
   * Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 30 mL/min according to the Cockcroft Gault formula
   * All premenopausal women and women within 12 months of menopause with a negative serum pregnancy test;
   * Left ventricular ejection fraction (LVEF) ≥ 50%;
   * Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy. Patients should be waited for at least 1 week to do the above tests if they have received thrombopoietin and/or granulocyte colony-stimulating factor.
9. Expected survival time of more than 6 months
10. Eligible patients of childbearing potential (men and women) must agree to use a reliable method of contraception (including intrauterine device, contraceptive or condom for females; condom or abstinence for males) with their partners prior to the study entry, during the trial, and for at least 180 days after completion of treatment. In addition, female patients should be non-lactating.
11. Patients must be informed of the study prior to the trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Patients who are known allergy or intolerance to investigational product, BCG or excipients.
2. Patients who have muscle-invasive bladder cancer (T2-T4) confirmed.
3. Patients who have concurrent extra-vesical (i.e., urethral, ureter or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium.
4. Patients who have a history of vesicoureteral reflux.
5. Patients who have not recovered from toxicity reactions associated with prior antitumor therapy except for fatigue and alopecia (determination criteria: toxicity remains > Grade 1 or has not returned to baseline levels).
6. Patients who have severe or uncontrollable cardiac diseases which need to be treated, including:

1). patients with severe arrhythmias (ventricular arrhythmias which requires clinical intervention, second to third degree of atrioventricular block, etc.); 2). patients with a medical history of myocardial infarction, unstable angina, angioplasty, or coronary artery bridging surgery within 6 months prior to the first dose of the investigational product; 3). patients with Class III or IV of congestive heart failure classified by NYHA 4). corrected QTc interval is > 450 ms for men and > 470 ms for women (calculated by the Fridericia formula) by 12-lead ECG at screening.

7. Patients who have received intravesical instillation therapy within 28 days prior to the first dose (patients are allowed to have immediate chemotherapeutic instillation in the past and after the current electrodesiccation); 8. Patients who have received antitumor therapy such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, biologic therapy and herbal medicine within 28 days or 5 half-lives of the drug (whichever is longer) prior to the first dose.

9. Patients who have participated in any other clinical trial (except for patients at overall survival follow-up) within 28 days or 5 half-lives of the drug (whichever is longer) prior to the first dose.

10. Patients who have additional malignancy that have had progression or requires active treatment in the last 3 years. Exceptions include, but are not limited to, in situ cervical cancer, superficial or non-invasive bladder cancer, basal cell carcinoma, in situ squamous cell carcinoma, or gastrointestinal tumors confined to the mucosal layer and that have been endoscopically resected.

11. Patients who have received allogeneic stem cell or solid organ transplantation.

12. Patients who have received any live/attenuated vaccine within 4 weeks or blood transfusion within 2 weeks prior to enrollment. 13. Patients who have received extensive radiotherapy to the pelvis (> 30% of the bone marrow area).

14. Patients who have an active autoimmune disease that have required systemic therapy in the past 2 years (i.e., with use of corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic therapy.

15. Patients who have a diagnosis of immunodeficiency or are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the planned first dose. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor.

16. Patients who have serious or poorly controlled disease, including but not limited to:

1. . active tuberculosis (with clinical signs, physical examination findings or radiographic findings of active tuberculosis);
2. . hepatitis B virus (HBV) infection with HBV DNA positive (>upper limit of detection values in the site), hepatitis C virus (HCV) infection with HCV RNA positive (>upper limit of detection values in the site), and human immunodeficiency virus (HIV) test positive;
3. . uncontrolled hypertension after treatment (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg);
4. . severe and uncontrollable pulmonary disease (severe infectious pneumonia, interstitial lung disease, etc.) (≥Grade 3, CTCAE);
5. . uncontrolled all types of serious infections (≥Grade 3, CTCAE), including active or refractory urinary tract infections.
6. . ascites, pleural effusion or pericardial effusion requiring drainage prior to first study drug therapy.

17. Patients with known history of psychiatric disorder, substance abuse, drug and alcohol use that would interfere with the subject's ability to cooperate with the requirements of the trial.

18. Patients who are inappropriate for participation in this trial in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-10-07 (Estimated); Study Completion 2026-12-07 (Estimated)

PRIMARY OUTCOMES:
DLTs occurrence | 21 days
  The DLT evaluation period is defined as 21 days after the first administration of investigational product.

SECONDARY OUTCOMES:
MTD | 21 days
  During DLT evaluation period, if ≥2 cases DLTs occur in the 3 or 6 subjects in one dose group, the previous dose is defined as MTD.

CONTACTS AND LOCATIONS:
Overall Officials: ye dingwei, M.D., Principal Investigator — Cancer Hospital affiliated to Fudan University